CLINICAL TRIAL: NCT05371756
Title: The Texas Immuno-Oncology Biorepository: Collection of Patients' Biospecimens for Analysis of Immunological and Molecular Biomarkers That Predict Benefit/Resistance to Cancer Therapeutics.
Brief Title: The TIOB - Collection of Patients' Biospecimens for Analysis of Immunological and Molecular Biomarkers.
Acronym: TIOB
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: Translational Genomics Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 019-350
Record Dates: First submitted 2022-04-27; First posted 2022-05-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: Biorepository; Immuno-Oncology; Molecular Biomarkers; Benefit & Resistance
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — TIOB will collect tissue, bodily fluids, and blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Texas Immuno-Oncology Biorepository (TIOB) is to collect and store well-defined and well-annotated serial biospecimens of tissue, blood, urine and stool in a longitudinal manner from cancer patients who are receiving either standard of care surgical interventions and or FDA approved immunotherapeutics across the largest not-for-profit health system in Texas. Comprehensive clinical and radiological data from a diverse population of patients with different racial, social and ethnic backgrounds matched with serial biospecimens over a patients journey with cancer marks the TIOB as a unique research facility.

DETAILED DESCRIPTION:
The goal of establishing the Texas Immuno-Oncology Biorepository (TIOB) is to create a research facility that purposely consents patients to collect, catalog, process, store, and analyze biospecimens with well-annotated clinical/radiological data from patients receiving surgical interventions or immunotherapeutics in our combined clinics throughout Texas. Potential types of studies that will be enabled by this resource will include but are not limited to (a) morphological studies including immunohistochemistry, (b) genomic and molecular analysis, including circulating, cell-free DNA, RNA, as well as extracellular vesicles and their cargo, (c) proteomic analysis involving protein isolation, (d) interrogation of circulating immune cells as well as the underlying tumor immune microenvironment, and (e) single-cell and spatial transcriptomics. Correlation of these studies with clinical, treatment outcome, and demographic information will be possible. Translation of multi-omics technologies will be a key feature of the TIOB and data integration strategies including genomics, epigenomics, transcriptomics, proteomics, radiomics, metabolomics and microbiomics will be possible and offer opportunities to improve our understanding of the complex biological interactions that define cancer.

ELIGIBILITY:
Inclusion Criteria:

* Understand and willingness to sign written informed consent method.
* Patients who are suspected by a physician of being at risk for developing cancer.
* Patients with confirmed or clinically suspected malignancy by a physician. This includes but is not limited to candidates for immunotherapy, surgical candidates, patients receiving Standard of Care drugs, immunotherapy drugs, participating on a clinical trial with immunotherapy drugs, patients who have received immunotherapy drugs in the past, patients with any other approved or investigational disease management.

Exclusion Criteria:

* Patients unwilling to donate blood
* Patients unwilling to provide informed consent for the collection of fresh or archived tumor tissue.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients due to receive or who have received immunotherapeutic drugs.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2050-09-11 (Estimated); Study Completion 2052-09-11 (Estimated)

PRIMARY OUTCOMES:
Develop a biorepository | 30 years
  Develop a biorepository that ensures molecular integrity and clinical relevance of quality human biospecimens and aligned clinical data for development of new diagnostic and therapeutic technology.
Release of specimens | 30 years
  Implement release of specimens from biorepository for testing.

SECONDARY OUTCOMES:
Laboratory Testing | 30 years
  Immunohistochemistry
Laboratory Testing | 30 years
  Genomic and Molecular analysis including circulating cell free DNA/RNA
Laboratory Testing | 30 years
  Proteomic analysis
Laboratory Testing | 30 years
  Single cell and Spatial transcriptomics

CONTACTS AND LOCATIONS:
Overall Officials: Ronan J Kelly, MD, MBA, Principal Investigator — Baylor Scott & White Research Institute
Locations (1):
- Baylor Scott & White Research Institute, Dallas, Texas, United States

REFERENCES:
- [Result] Yehonatan Elon et al. Longitudinal plasma proteomic analysis: A monitoring strategy for NSCLC patients treated with immunotherapy.. J Clin Oncol 43, 8579-8579(2025). DOI:10.1200/JCO.2025.43.16_suppl.8579
- [Result] Kelly RJ, Whitsett TG, Snipes GJ, Dobin SM, Finholt J, Settele N, Priest EL, Youens K, Wallace LB, Schwartz G, Wong L, Henderson SM, Gowan AC, Fonkem E, Juarez MI, Murray CE, Wu J, Van Keuren-Jensen K, Pirrotte P, Highlander S, Contente T, Baker A, Victorino J, Berens ME. The Texas Immuno-Oncology Biorepository, a statewide biospecimen collection and clinical informatics system to enable longitudinal tumor and immune profiling. Proc (Bayl Univ Med Cent). 2022 Aug 26;36(1):1-7. doi: 10.1080/08998280.2022.2114129. eCollection 2023. PMID 36578607

DOCUMENTS (1):
  • Informed Consent Form (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT05371756/ICF_000.pdf